CLINICAL TRIAL: NCT06957977
Title: A Randomized Controlled Study of Endoscopic Cryoablation Combined With PD-1 Inhibitor for Maintenance Therapy in Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhongguang Luo, MD (Other)
Responsible Party: Sponsor-Investigator, Zhongguang Luo, MD, Chief Physician, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-081
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer; Cryoballoon Ablation
Keywords: Cryoballoon ablation; ECAT; PD-1
MeSH Terms: conditions — Stomach Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: Patients will first receive standard treatment regimens (such as FOLFOX, POLF, FLOT, SOX, CAPOX, or FOLFIRI). Among these, 30 patients with advanced gastric cancer who achieve a partial response (PR) following standard treatment will undergo peripheral blood and local tumor tissue immunological evaluations, and will then be randomly assigned into two groups. Twenty patients will receive gastric local endoscopic cryoballoon ablation treatment (ECAT) combined with sintilimab, while ten patients will receive sintilimab monotherapy. Subsequently, both groups will continue with standard maintenance therapy, followed by assessments of treatment efficacy and safety.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECAT + PD-1 (Experimental): Patients who achieve a partial response (PR) following standard treatment will subsequently receive gastric local endoscopic cryoballoon ablation treatment (ECAT) combined with sintilimab. Sintilimab will be administered within three days before and after the ECAT procedure, and continued regularly thereafter.
  Interventions: Procedure: Endoscopic Cryoballoon Ablation Treatment; Drug: PD1 Inhibitor
- PD-1 (Active Comparator): The remaining 10 patients who achieve a partial response (PR) following standard treatment will receive sintilimab monotherapy, followed by standard maintenance therapy.
  Interventions: Drug: PD1 Inhibitor

INTERVENTIONS:
Procedure: Endoscopic Cryoballoon Ablation Treatment — ECAT: A cryoballoon with catheter is inserted along the endoscopic forceps channel, the balloon is placed on the surface of the tumor, and the balloon is dilated so that it fits snugly over the lesion. The freezing cycle is initiated and continued for 2-3 minutes, and then the balloon is rewarmed and frozen again for 2-3 minutes; the freeze-rewarm cycle is repeated twice. PD-1:The first PD-1 monoclonal antibody treatment in this study was given within 3 days before and after ECAT treatment, and subsequent treatment was given every three weeks according to the instructions.
  Other Names: ECAT
  Arms: ECAT + PD-1
Drug: PD1 Inhibitor — The first administration of the PD-1 monoclonal antibody is initiated when patients achieve a partial response (PR) following standard treatment. Subsequent administrations are given every three weeks according to the prescribing information.

SUMMARY:
This study evaluates the safety and efficacy of endoscopic cryoballoon ablation treatment (ECAT) combined with a PD-1 inhibitor (sintilimab) as maintenance therapy in patients with advanced gastric cancer, and further explores the underlying immunoregulatory mechanisms.

DETAILED DESCRIPTION:
This study is a single-center, randomized, controlled, open-label, prospective clinical trial. A total of 42 patients with advanced gastric cancer will be enrolled. Among them, 30 patients who achieve a partial response (PR) after receiving standard of care (SOC) treatment - such as FOLFOX, POLF, FLOT, SOX, CAPOX, or FOLFIRI - will be randomly assigned to two groups. Twenty patients will receive local gastric endoscopic cryoballoon ablation treatment (ECAT) combined with sintilimab, while the remaining ten patients will receive sintilimab monotherapy. Both groups will subsequently undergo standard maintenance therapy, followed by assessments of treatment efficacy, safety, and immunological evaluations of both peripheral blood and tumor tissues. Patients whose disease status is assessed as stable disease (SD) or progressive disease (PD) after SOC treatment will proceed to receive standard second-line therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with advanced gastric cancer (stage IV according to the AJCC 8th edition, including locally advanced unresectable gastric cancer [stage IVa] and gastric cancer with distant metastasis [stage IVb]; Borrmann classification types I, II, or III) who are deemed ineligible for surgical resection or unable to tolerate surgery, and meet the indications for first-line therapy with sintilimab combined with fluoropyrimidine- and platinum-based chemotherapy;
2. Age ≥18 years;
3. WHO pathological types: adenocarcinoma or neuroendocrine tumors;
4. Physician-assessed estimated life expectancy greater than 3 months, with distant metastases considered controllable;
5. Maximum diameter of the primary tumor ≤6 cm;
6. Adequate major organ function, defined as:① Liver function: ALT and AST ≤ 2.5 times the positive range, total bilirubin ≤ 2.0mg/dL; ② Renal function: creatinine clearance ≥ 40mL/min calculated using the EPI formula;
7. Hematological criteria: hemoglobin (Hgb) ≥70 g/L; absolute neutrophil count (ANC) ≥1.5×10⁹/L; platelet count (PLT) ≥80×10⁹/L;
8. Coagulation function: prothrombin time (PT) and activated partial thromboplastin time (APTT) both <2 times the normal value;
9. Negative pregnancy test for women of childbearing potential;
10. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
11. Signed informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women planning to become pregnant within six months;
2. Patients with infectious diseases (such as HIV, syphilis, or active tuberculosis);
3. Patients with active hepatitis B or hepatitis C infection;
4. Patients with other concurrent primary malignancies;
5. Patients who have participated in another clinical trial within the past month;
6. Patients who have taken antiplatelet or anticoagulant medications within the past week;
7. Patients with gastric cancer complicated by active bleeding;
8. Patients with massive ascites (ascites volume ≥3000 mL);
9. Patients with cardia obstruction or pyloric obstruction;
10. Patients with active infections or autoimmune diseases;
11. Patients deemed unsuitable for treatment by the investigator for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to study completion, assessed up to 2 years
  PFS is measured from the start of treatment until the first documented evidence of disease progression (based on RECIST 1.1) or death from any cause, whichever occurs first.
Overall-Survival (OS) | From enrollment to study completion, assessed up to 5 years
  The length of time from the start of treatment until death from any cause.

SECONDARY OUTCOMES:
Percentage of participants achieving complete remission (CR) and partial remission (PR) after treatment | 3 to 24 weeks after the end of treatment
  Objective remission rate (ORR), the percentage of participants whose tumors shrink by a certain amount and remain there for a certain period of time, including complete remission (CR) and partial remission (PR). CR (Complete remission): Complete disappearance of the target lesion, with no new lesions produced, and lasting for more than 4 weeks. PR (Partial remission): the sum of the largest diameters of the target lesions is reduced by more than 30%, and lasts for more than 4 weeks.
Percentage of participants achieving remission (PR+CR) and lesion stabilization (SD) after treatment | 3 to 24 weeks after the end of treatment
  Disease control rate (DCR) is the percentage of participants who achieve remission (PR+CR) and stabilization of lesions (SD) after the treatment. Stable disease (SD) means that the sum of the largest diameters of the tumor lesions has not shrunk to PR, or has not enlarged to PD.
Number of participants with treatment-related adverse events | From the start of treatment to 24 weeks after the end of treatment
  The number of patients who experience ECAT-related adverse events (such as intraoperative bleeding, intraoperative perforation, postoperative bleeding, etc.)

OTHER OUTCOMES:
Number of immune cells in peripheral blood | From enrollment to study completion, assessed up to 24 weeks
  Peripheral blood will be analyzed for the number of immune cells after applying flow cytometry and mRNA sequencing.
Number of immune cells in tumor tissues | From enrollment to study completion, assessed up to 24 weeks
  Apply mRNA sequencing, immunohistochemistry and immunofluorescence to analyze the number of immune cells in tumor tissues, including CTL, Treg, DC, TAM, MDSC, NK, NKT and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai, Shanghai Municipality, China